CLINICAL TRIAL: NCT06405464
Title: Cabotegravir Plus Rilpivirine Long-acting Regimen in the Swiss HIV Cohort Study: Uptake, Outcome, and Risk Factors for Treatment Failures in a Real-world Setting
Brief Title: Cabotegravir Plus Rilpivirine Long-acting Regimen in the Swiss HIV Cohort Study:Uptake, Outcome, and Risk Factors for Treatment Failures
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss HIV Cohort Study (Network)
Responsible Party: Sponsor
Other Study IDs: 903_SHCS; 222485 (Other Grant/Funding Number: ViiV Healthcare)
Record Dates: First submitted 2024-04-15; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Tablets; Rilpivirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood (plasma and cell samples)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Swiss HIV Cohort Study participants on CAB+RPV LA regimen: Swiss HIV Cohort Study participants initiating the CAB+RPV LA regimen
  Interventions: Drug: VOCABRIA 30Mg Tablet; Drug: EDURANT 25Mg Tablet; Drug: Cabotegravir Injectable Suspension; Drug: Rilpivirine Injectable Suspension; Biological: Intact proviral DNA assay; Biological: Full-length sequencing
- Swiss HIV Cohort Study participants on a standard of care oral regimen: Matched control population on a standard of care oral regimen
  Interventions: Biological: Intact proviral DNA assay; Biological: Full-length sequencing

INTERVENTIONS:
Drug: VOCABRIA 30Mg Tablet — CAB 30 mg Film-coated tablets
  Other Names: Cabotegravir Tablets
  Groups: Swiss HIV Cohort Study participants on CAB+RPV LA regimen
Drug: EDURANT 25Mg Tablet — RPV 25 mg film-coated tablets
  Other Names: Rilpivirine Tablets
  Groups: Swiss HIV Cohort Study participants on CAB+RPV LA regimen
Drug: Cabotegravir Injectable Suspension — CAB LA 600 mg prolonged release suspension for injection (3 mL)
  Other Names: Vocabria
  Groups: Swiss HIV Cohort Study participants on CAB+RPV LA regimen
Drug: Rilpivirine Injectable Suspension — RPV LA 900 mg prolonged release suspension for injection (3 mL)
  Other Names: Rekambys
  Groups: Swiss HIV Cohort Study participants on CAB+RPV LA regimen
Biological: Intact proviral DNA assay — HIV-1 latent reservoir size
Biological: Full-length sequencing — Proviral DNA

SUMMARY:
This study aims to characterize Swiss HIV Cohort Study participants initiating the CAB+RPV LA regimen, assess adherence to Swiss label indications, and describe treatment outcomes in this large, multicentre, heterogeneous, high-income setting. Moreover, the study aims to assess virological, immunological, demographic, clinical, and behavioural factors associated with viral failure under CAB+RPV LA regimen.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the SHCS
* All SHCS participants initiating the CAB+RPV LA regimen
* All SHCS participants on SOC oral regimen

Exclusion Criteria:

* Not participating in the SHCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of SHCS participants initiating the CAB+RPV LA regimen and a matched control population on a SOC oral regimen (including dual drug regimens)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals with viral blips | Month 24
  Proportion of individuals with viral blips (defined as one HIV-1 RNA >50 and <400 c/mL with a next HIV-1 RNA <50 copies/ml)
Proportion of individuals with confirmed viral failures | Month 24
  Proportion of individuals with confirmed viral failures (defined as two consecutive HIV-1 RNA ≥ 50 c/mL)
Proportion of individuals switching off CAB+RPV LA to previous or another oral regimen | Month 24
  Proportion of individuals switching off CAB+RPV LA to previous or another oral regimen after HIV-1 RNA levels of >50 to <400 copies/mL and >400 copies/mL
Time to viral failure | Up to month 24
  Overall time to confirmed viral failures (defined as two consecutive HIV-1 RNA ≥ 50 c/mL)
Proportion of participants who discontinue treatment due to drug-related reasons | Month 24
  Proportion of participants who discontinue treatment due drug-related reasons and re-suppression regimens (such as adverse events, confirmed viral failure, low level viremia or low blood concentration measurements) including the choice of re-suppression regimens.
Proportion of participants who discontinue treatment due to drug-unrelated reasons | Month 24
  Proportion of participants who discontinue treatment due drug-unrelated reasons and re-suppression regimens (such as patient wish, death, migration, and loss to follow-up) including the choice of re-suppression regimens.
Proportion of participants by characteristics | Month 24
  - Proportion of participants by socio-demographic and clinical characteristic(s) (e.g., by age, sex, body mass index, race, geographic origin, education, transmission mode, HIV-1 RNA levels, CD4 cell count, duration of HIV-1 infection, HIV-1 subtype, previous regimen, genotypic resistance profile, coinfections, lifestyle variables, and co-medications)
Overall adherence to Swiss label indication in CAB+RPV LA prescriptions | Month 24
  - Overall adherence to Swiss label indication in CAB+RPV LA prescriptions between care providers, such as university hospital versus private physicians, and among nationwide centres
Overall adherence to the proposed injection schedules | Month 24
  - Overall adherence to the proposed injection schedules quantified by deriving an CAB+RPV LA adherence threshold (e.g., accounting for any missed injection, daily oral bridging ART, and delayed injection of +7 days according to the Swiss label indication)
Proportion of participants by treatment adherence category | Month 24
  - Proportion of participants by treatment adherence categories (e.g., optimal, sub-optimal, and poor adherence)

SECONDARY OUTCOMES:
Investigate in-depth factors associated with viral blips and viral failure | Month 24
  Proportion of individuals by risk factor(s) (e.g., by body mass index, race, geographic origin, education, HIV-1 RNA levels, CD4 cell count, duration of HIV-1 infection, HIV-1 subtype, previous regimen, treatment adherence, CAB+RPV LA plasma concentrations measured at time of failure, genotypic resistance profile , lifestyle variables, and co-medications)
Measure intact proviral DNA as potential predictor for viral failure | Month 24
  Measure intact proviral DNA as potential predictor for viral failure among PWH initiating CAB+RPV LA regimen and compare with the matched control population on a SOC oral regimen
Assessment of resistance associated mutations from proviral DNA as potential predictor for viral failure | Month 24
  Assessment of resistance associated mutations from proviral DNA as potential predictor for viral failure among PWH initiating CAB+RPV LA regimen and compare with the matched control population on a SOC oral regimen

CONTACTS AND LOCATIONS:
Overall Officials: Jessy J Duran Ramirez, MSc, Principal Investigator — Department of Infectious Diseases and Hospital Epidemiology, University Hospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided